CLINICAL TRIAL: NCT04322578
Title: Crizotinb or Standard Chemotherapy in Met Exon 14 Skipping Advanced Non-small Cell Lung Cancer
Brief Title: Crizotinb or Standard Chemotherapy in Met Exon 14 Skipping Advanced NSCLC
Acronym: CONFIRM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, professor, Hunan Province Tumor Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20203017
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Non-small Cell Lung Cancer
Keywords: non-small cell lung cancer; Crizotinb; Chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Crizotinib; 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine; Pemetrexed; Immune Checkpoint Inhibitors; Carboplatin; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A: Target Therapy Group. (Experimental): Patients with MET exon 14 skipping will be treated with First line crizotinib or savolitinib and other MET TKIs.
  Interventions: Drug: Crizotinib
- Cohort B: Chemotherapy or Chemotherapy plus immune checkpoint inhibitor (Experimental): Patients with MET exon 14 skipping will be treated with chemotherapy.
  Interventions: Drug: Pemetrexed

INTERVENTIONS:
Drug: Crizotinib — Crizotinib 250mg po bid. Savolitinib 300mg po, qd.
  Other Names: Savolitinib
  Arms: Cohort A: Target Therapy Group.
Drug: Pemetrexed — Pemetrexed, 500mg/m2, ivgtt erery 21day.
  Other Names: immune checkpoint inhibitors; Carboplatin; Bevacizumab
  Arms: Cohort B: Chemotherapy or Chemotherapy plus immune checkpoint inhibitor

SUMMARY:
This study aims to explore the efficacy and safety of Crizotinb or Standard Chemotherapy in Met exon 14 skipping Advanced Non-small Cell Lung Cancer

DETAILED DESCRIPTION:
This study aims to explore the efficacy and safety of Crizotinb or Standard Chemotherapy in Met exon 14 skipping Advanced Non-small Cell Lung Cancer . All the clinical and survival data will be collected for full analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Understand the requirements and contents of the clinical trial, and provide a signed and dated informed consent form.
2. Age ≥ 18 years.
3. Histopathology or cytology confirmed and recorded local progression or metastatic non-small cell lung cancer without systemic treatment.
4. MET exon 14 skippign confirmed by an accredited local laboratory.
5. ECOG 0 - 1.
6. Predicted survival ≥ 12 weeks.
7. Adequate bone marrow hematopoiesis and organ function
8. Presence of measurable lesions according to RECIST 1.1.
9. Subjects with stable brain metastases may be included in the study.

Exclusion Criteria:

1. Prior systemic therapy for locally advanced or metastatic disease.
2. Subjects who have received any of the following treatments must be excluded:

   * Treatment with molecules such as EGFR, VEGFR antibodies within 4 weeks prior to the first dose of study drug.
   * Have received radiation within 14 days prior to the first dose or have not recovered from radiation-related toxicity. Chest and extra-brain palliative radiotherapy, stereotactic radiosurgery, and stereotactic body radiotherapy may be performed 7 days prior to the first dose.
   * Ongoing (or inability to discontinue) possibly potent CYP1A2, CYP3A inhibitor (1 week), or inducer (2 weeks) drug therapy or herbal supplements within 1-2 weeks prior to the first dose.
3. Presence of spinal cord compression or meningeal metastasis.
4. History of other malignant tumors within 2 years.
5. Adverse events (except alopecia of any degree) of CTCAE > grade 1 due to prior treatment (e.g., adjuvant chemotherapy, radiotherapy, etc.) prior to the first dose.
6. History of stroke or intracranial hemorrhage within 6 months prior to the first dose.
7. The presence of any severe or poorly controlled systemic disease, including poorly controlled hypertension and active bleeding in the judgment of the investigator.
8. Subjects with persistent or active infection, including but not limited to hepatitis B (HBV), hepatitis C (HCV), human immunodeficiency virus (HIV) and COVID-19 infection.
9. Heart-related diseases or abnormalities
10. Past history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis requiring steroid therapy or interstitial lung disease with active clinical symptoms, immune pneumonia caused by immunotherapy.
11. Refractory nausea and vomiting, chronic gastrointestinal disease, difficulty swallowing drugs, or inability to adequately absorb sunvozertinib or anlotinib due to previous bowel resection.
12. Live vaccine was given 2 weeks before the first medication.
13. Women who are breastfeeding or pregnant.
14. Hypersensitivity to the test drug and the ingredients.
15. Other conditions assessed by the investigator to be unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-03-24 (Actual); Primary Completion 2025-03-24 (Estimated); Study Completion 2026-03-24 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Time from first subject dose to study completion, or up to 36 month
  PFS defines as first dose to first documented disease progression assessed by investigator or death due to any cause

SECONDARY OUTCOMES:
Overall survival (OS) | Time from first subject dose to study completion, or up to 36 month
  To assess overall survival, define as first dose to the death of the subject due to any cause
Objective Response Rate (ORR) | Time from first subject dose to study completion, or up to 36 month
  To assess Chemotherapy and TKIs overall response rate according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by investigator, define as the proportion of subjects who have a complete response (CR) or a partial response (PR)

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Zhang, MD, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Yongchang Zhang, Changsha, Hunan, China